CLINICAL TRIAL: NCT04693364
Title: 3D Printed Breast Models: Acceptability of Personalized Models in Breast Cancer Patients
Brief Title: Acceptability of 3D Printed Breast Models as Surgical Decision Aids for Breast Cancer Treatment
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0817; NCI-2020-13314 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0817 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaire, 3D breast model, discussion): Patients complete questionnaire over 5 minutes about difficulties in making decision about breast cancer treatment, then participate in a consultation with regular care doctor and study doctor/study staff using the 3D breast model. Patients then complete questionnaires over 5-10 minutes about their opinions on the breast model and different breast surgical treatment options available.
  Interventions: Other: Decision Aid; Procedure: Discussion; Other: Questionnaire Administration

INTERVENTIONS:
Other: Decision Aid — Use 3D printed breast model
Procedure: Discussion — Participate in consultation
  Other Names: Discuss
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study is to find out the acceptability of a 3D printed breast model by patients as they consider their surgical treatment options. Researchers also want to learn the possible impact of the 3D printed breast model in the patient's decision making process.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine feasibility and explore the acceptability of 3 dimensional (3D) printed breast models as a decision aid in breast cancer treatment decision making.

OUTLINE:

Patients complete questionnaire over 5 minutes about difficulties in making decision about breast cancer treatment, then participate in a consultation with regular care doctor and study doctor/study staff using the 3D breast model. Patients then complete questionnaires over 5-10 minutes about their opinions on the breast model and different breast surgical treatment options available.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Women diagnosed with breast cancer
* Patient is a candidate for surgical management
* Patient has a surgeon at MD Anderson Cancer Center (MDACC) (main campus and/or regional care centers) who has agreed to have the 3D model created
* Patients with a breast magnetic resonance imaging (MRI) performed at the MD Anderson (at the West Houston location as well as main campus)
* Patient able to speak, read or write English
* PHYSICIAN ELIGIBILITY: Breast surgeon

Exclusion Criteria:

* Pregnant and breast feeding patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer who are candidates for surgical management and agreed to have a 3D model created
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Change in patient decisional conflict | 45 minutes - up to 12 months
  Will be assessed based on changes in decisional conflict scale data collected before and after use of the 3 dimensional (3D) printed breast model during consultation with the breast surgeon using paired sample t-tests.
Acceptability of the 3D model | 45 minutes - up to 12 months
  Will be measured with questions adapted from the Ottawa measures. 'Acceptability' (of a decision aid) refers to ratings regarding the comprehensibility of components of a decision aid, its length, pace (if audio-visual), amount of information, balance in presentation of information about options, and overall suitability for decision making. Responses are reported descriptively in terms of the proportions of patients responding positively or negatively on each criterion.

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Arribas, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MDAndersonCancerCenterWebsite — http://www.mdanderson.org